CLINICAL TRIAL: NCT03067779
Title: Is There a Digital Divide in Chronic Kidney Disease (CKD)?
Acronym: eCRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Pennsylvania (Other); University of Maryland (Other); University of Illinois at Chicago (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00057833
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey and mHealth Tool (Other): A survey has been designed that evaluates CRIC participants' computer and mobile phone usage, and perceived e-health literacy.
  There is also a mobile health-based (mHealth) patient safety educational curriculum that evaluates CRIC participants' knowledge of patient safety hazards in CKD. The mHealth patient safety curriculum tool is also known as eCRIC.
  Interventions: Other: mHealth Tool

INTERVENTIONS:
Other: mHealth Tool — The curriculum in the mHealth tool was derived in consultation with patient safety, informatics and adult educational curricula experts, and is comprised of clinical vignettes describing common patient safety themes in CKD and includes a pre- and post-test knowledge assessment. Topics of emphasis included NSAID risk awareness, hypoglycemia awareness, avoidance of volume depletion when ill ("Sick Day Protocol") and avoidance of contrast-induced nephropathy.

SUMMARY:
This study is looking to improve the safety of patients with chronic kidney disease via education provided on a mobile tablet. This study will additionally examine if electronic tools, such as mobile tablets, can help.

DETAILED DESCRIPTION:
Individuals with CKD are at risk for adverse safety events, yet little is known regarding the utility of health information technology (IT) educational tools to reduce these events. The results of this project will be invaluable in gaining a better understanding of the limitations and potential for use of a patient-centered mHealth patient safety educational intervention in high-risk individuals with CKD.

The study will evaluate the perceived eHealth literacy of patients with CKD and its relation to medication errors in the CRIC cohort. The hypothesis is that a novel mHealth-based patient safety curriculum designed to address a wide-range of e-literacy will be effective in attenuating the identified Digital Divide adversely affecting many CKD patients, and will reduce adverse safety events common in this population.

Study Aims:

1. Examine the association between surveyed perceived e-literacy and medication errors in individuals with CKD

   Hypothesis 1: Medication error rates will be higher among CRIC participants with low eHealth literacy.
2. Assess the acceptance and feasibility of a novel mHealth-based patient safety curriculum to improve patient safety risk knowledge among individuals with CKD and determine its efficacy in increasing patient safety risk awareness.

Hypothesis 2a: A low literacy mHealth patient safety curriculum will improve patient safety risk awareness among high risk individuals with CKD.

Hypothesis 2b: Medication error rates will be higher among CRIC participants with low patient safety risk awareness.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Chronic Renal Insufficiency Cohort (CRIC) Study.

Exclusion Criteria:

* Not enrolled in Chronic Renal Insufficiency Cohort (CRIC) Study.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Medication Errors | 10 minutes
  eHealth Literacy questionnaire and how that relates to medication errors
e-literacy questionnaire | 10 minutes
  eHEALS portion of the questionnaire will be used to determine eHealth literacy and e-literacy

SECONDARY OUTCOMES:
Patient Safety Risk | 20 minutes
  mHealth tool and how that relates to patient safety risk

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa J Diamantidis, MD, MHS, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University School of Medicine, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The research team will not be sharing IPD with other researchers.